CLINICAL TRIAL: NCT06953622
Title: Establishment of a Clinical and Prognostic Follow-up Cohort of Migraine Patients With Patent Foramen Ovale
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024296
Record Dates: First submitted 2024-08-19; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-07

CONDITIONS: Migraine; Patent Foramen Ovale
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Conservative group: Don't use antiplatelet drugs or undergo patent foramen ovale closure.
  Interventions: Drug: Conservative treatment
- Antiplatelet group: The application of antiplatelet drug.
  Interventions: Drug: Antipaletet drug
- PFO group: Receive a patent foramen ovale closure surgery.
  Interventions: Procedure: Patent Foramen Ovale Closure

INTERVENTIONS:
Drug: Conservative treatment — Receive no antipaletet drug treatment and surgery
  Groups: Conservative group
Drug: Antipaletet drug — Use of antipaletet drugs.
  Groups: Antiplatelet group
Procedure: Patent Foramen Ovale Closure — Receive the surgery of Patent Foramen Ovale
  Groups: PFO group

SUMMARY:
To establish a headache center in China that combines clinical, imaging and laboratory examinations, explore the feasible treatment options for migraine combined with patent foramen ovale, and search for the possible influencing factors, construct models that influence prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for migraine in the International Classification of Headache (ICHD-3);
* Confirmation of patent foramen ovale through transthoracic echocardiography(TTE) or transesophageal echocardiography(TEE)/right heart contrast echocardiography
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Can not sign the informed consent form or cooperate with follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All clinically confirmed migraine patients with PFO who met the inclusion criteria were included.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of migraine attacks | 3 months, 6 months, 1 year, 2 years and 3 years
  Migraine attacks are an important indicator of improvement in symptoms. The comparison measures included headache frequency, duration, pain degree, VAS scores, HIT-6 scores, HAMA, HAMD, and PSQI.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China